CLINICAL TRIAL: NCT06243861
Title: Attachment Bonding and Neonatal Hospitalization: the Impact of Hospitalization in a Kangaroo Unit
Acronym: UKLA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-08Obs-CHRMT
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Postnatal Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- kangaroo unit
  Interventions: Behavioral: Mother-child bond
- postnatal care
  Interventions: Behavioral: Mother-child bond

INTERVENTIONS:
Behavioral: Mother-child bond — assessing whether the mother-child bond is degraded in the UK, in comparison with that of mothers in post-natal care

SUMMARY:
The Kangaroo Unit (UK) takes care of newborns requiring special care or monitoring for a pathology whose clinical situation is stable and whose prognosis is favorable. In order to avoid separating mother and child, these units were created with a care pathway somewhere between that requiring hospitalization in a neonatal unit and that of pathology-free newborns in post-natal care. Theoretically, the mother-child bond created in the UK is as good as that created in conventional post-natal care. However, studies show that there are limits to the quality of the bond in the UK. This study aims to assess whether the mother-child bond is degraded in the UK, in comparison with that of mothers in post-natal care.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age, hospitalized in a Kangaroo Unit or in a post-natal unit,
* Affiliated to a social security scheme,
* fluent in French
* no objection of participation

Exclusion Criteria:

* Patient who :

  * given birth to a child who was stillborn or died at birth
  * difficulty understanding written French
  * psychological incapacity (psychiatric disorder, too great a vulnerability) or physical incapacity (physical/motor disability) to answer questionnaires,
* Patient under court protection, guardianship or curatorship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — study conducted in mothers
Study Population: patient hospitalized in a Kangaroo Unit or in a post-natal unit
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Mother-infant bonding | Up to 3 days after delivery
  Mother-infant bonding score from Taylor's Mother to Infant Bonding Scale (MIBS)

SECONDARY OUTCOMES:
Assessment of mothers' state and trait anxiety levels | Up to 3 days after delivery
  using Spielberger's STAY form Y1 and Y2: a self-reported questionnaire with 20 items assessed on a 4 points scale
Assessment of perceived parenting competence | Up to 3 days after delivery
  using Gibaud-Wallston's Parenting Sense of Competence Scale (PSOC). The PSOC is a 17 item scale, with 2 subscales. Each item is rated on a 6 point Likert scale anchored by 1 = "Strongly Disagree" and 6 = "Strongly Agree".
Assessment of patients' quality of life | Up to 3 days after delivery
  using the McGill Quality of Life Questionnaire (MQOL). consists of 14 items divided into four domains: The Single-Item Scale (SIS), physical symptoms (three items), feelings and thoughts (seven items), and social (three items).

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure BOYE, Principal Investigator — CHR Metz Thionville
Locations (1):
- CHR Metz-Thionville/Hopital Mercy, Metz, France

IPD SHARING:
Plan to Share IPD: No